CLINICAL TRIAL: NCT04157439
Title: Compare the Effects of Two Manual Treatment Regimens on Individuals With Upper Trapezius Trigger Points
Brief Title: Manual Treatment Regimens in Upper Trapezius Trigger Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Shiza Sultan-REC00382
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Integrated Neuromuscular Inhibition Technique; Muscle Energy Technique; Neck Disability Index
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Hot fermentation, Sustain pressure on trigger point, Self-stretches
  Interventions: Other: Control Group
- Experimental Group (Experimental): Integrated Neuromuscular Inhibition Technique Post isometric stretch (MET) Strain counter strain
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Control Group — Hot fermentation was applied for 10 mints Sustain pressure on trigger point was applied with thumb for 3secs hold and 2 sec release (till pain is reduced).
  Self-stretches of cervical muscles (10 reps× 1set) For home plan cervical muscles stretching and postural care was guided
  Arms: Control Group
Other: Experimental Group — Hot fermentation was applied for 10 mints. Integrated Neuromuscular Inhibition Technique [sustain pressure, Post Isometric Relaxation (PIR) and SCS]. Sustain pressure was applied on trigger points using thumb for 3 sec hold and 2 mints release (till pain is reduced).
  Post isometric stretch (MET) was given with 4 repetitions (6-10sec hold). Strain counter strain was given in which upper trapezius shortened position was maintained by slight flexion, same side bending, opposite rotation and shoulder abduction for 90 sec and repeats this procedure till the pain is reduced to 3 out of 10.
  Self-stretches for cervical muscles were done at the end of session to maintain the gained ranges (10 reps×1 set) For home plan cervical muscles stretching and postural care was guided
  Arms: Experimental Group

SUMMARY:
To compare the effect of sustain pressure and Integrated Neuromuscular Inhibition Technique on individuals with upper trapezius Trigger points (TrPs). The Study Design was Randomized control trial. According to inclusive criteria 26 patients were randomly allocated by sealed envelope method in experimental and control group. Patients were assessed at baseline and 4th day of session on NPRS, NDI questionnaire and ranges were taken by Goniometer and pressure threshold by Algometer. There was 3 drop out and the reason was loss of follow up. Hot pack was applied to both groups for 10mints before session. Sustain pressure was given for 3sec hold and 2sec release till pain decreases in control group. While, in experimental group INIT was used. Sustain pressure was applied on MTrPs for 3sec hold and 2sec release till pain decreases, Post isometric relaxation (MET) was given with 6-10 sec hold and repeat 4 times and at last Strain counter-strain (SCS) was given to hold muscle in shortest position for 90sec or pain reduced to 3 out of 10. At last cervical stretches were given and home plan was guided.

DETAILED DESCRIPTION:
In clinical practice the neck and head pain is the most shared problem throughout the population. 45% to 54% of the total population is affected by neck pain. Idiopathic neck prevalence during lifetime is approximately 67% to 71%, two third of whole population will experience some event of neck and head pain in some stage of their life. One of important health problem is headache which is increasing mechanism of these disorders. 38.3% population experienced tension type headache in a studies during 1 year and out of which 2.2% had the chronic cases. Occurrence of cervicogenic headache in a Scandinavian individuals was nearly 16%. In recent years other studies done on general population the estimated percentage of migraine experienced by adults was 10% to 12%. And prevalence of other type of headaches is increased tremendously in past few years. Work and activity which is limited due to this disability was documented by 60% of patients having headache. 64% working capacity was reduced because of headache. So, it is important that headache has reduced the quality of life generally Trigger point are very common but still they are overviewed and poorly managed due to practitioners who have less information regarding management of trigger points. Since long time practitioners have acknowledged the management of painful and tender muscles by stretching or elongating its fibers. Muscles having trigger points are tense when examined and it has also restricted ranges. This exaggerated tension in muscle is misinterpreted with muscle spasm

* Trigger point pain is unique and tender point in skeletal muscle or fascia that does not occur due to injury, degenerative changes, malignancy, acute infection and others.
* On palpation trigger point is like a taut band, knot or a bump under the finger in a muscle which produces a local twitch response on activation.
* When trigger point is compressed the patient reports pain in a specific pattern and give jump sign.

Clinical diagnosis presents with local tenderness and 'jump sign' due to hyperirritability of the taut band, but still it is not known that if MTrPs is due to joint and bone problem or it is a separate disorder. Current studies have theorized that pathophysiology of myofascial pain syndrome and the creation of trigger points are due to damaged or burdened muscle threads, which results in automatic shortening and decreased supply of oxygen and nutrient, and with greater metabolic demand on local tissues. While the lengthened muscle have different pathophysiology for activating MTrPs. It is also suggested that reduced elasticity of neural structures is due to decrease in length of upper trapezius muscle Referred pain pattern and location of central trigger point 1 in the middle of vertical fibers of upper part of trap muscle. The central trigger point 2 in the middle of the horizontal fibers of the upper part of the trapezius. Central point 3 is in lower fibers of trapezius muscle. Trigger point 4 is at the lateral attachment of the lower fibers of trapezius muscle. This painful area is enthesopathy at the end of the tight bands associated with trigger point 3. In middle fibers of trapezius trigger point 5 is found, whereas 6th trigger point is found at the lateral attachment of middle fibers. The trigger point 7 is also in middle fibers Sustain pressure is application of gradually strong, painful pressure on trigger point for management of trigger points. By applying progressive pressure the ischemia is produced at local point using thumb or pressure Algometer and gradually the pain is reduced thus the investigators increase the pressure and it should be followed by increasing the length of the shortened muscle Muscle energy technique (MET) is a manual procedure in which minimal energy is used for management of movement limitation in spine and extremities. Osteopathic MET is a unique procedure conventionally used to treat muscular tension, local edema, empty end feel and joint dysfunction. For achieving good results in MET co-ordination of patient and therapist is required, whereas patient actively participate by contracting his/her muscles actively. It defined MET as a manual method in which patient contracts actively against the opposing force applied by the therapist. MET is used for management of shortened, stiffened or tightened muscles fibers. It is also used to strengthened the weak muscles.

Myofascial pain is managed better when treatment is applied at the specific point i.e. MTrPs there are many methods used manually for management of trigger points some of them are sustain pressure, MET, positional release technique and Integrated neuromuscular inhibition technique (INIT). Combined MET, sustain pressure and strain counter strain for the better management of the trigger points and it is known as integrated neuromuscular inhibition technique and its effect can be obtained by using multidimensional methodology Sustain pressure is most commonly used for the management of trigger points in clinical setups. The purpose of my study is to use INIT for the management of trigger points, in this technique the investigators apply sustain pressure along with muscle energy technique post isometric relaxation and Strain counter strain. After the sustain pressure it was necessary to stretch and lengthen the muscles so the reoccurrence of trigger point will be minimize. The strain counter strain normalized the sensory abnormal input to normal input and through this the investigators also minimize the chance of reoccurrence of trigger point. The significance of the study is to increase the quality of care that consequences the independent life

ELIGIBILITY:
Inclusion Criteria:

* Limited range of motion (ROM): side bending or rotation (any side)
* Pain more than 3 on NPRS
* Upper trapezius triggers points: any one

Exclusion Criteria:

* Radiculopathies
* Malignancy
* Infection
* Trauma
* Positive vertebrobasilar insufficiency (VBI)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-08 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 4th day
  Changes from the baseline, NDI consist of 10 items that are pain, personal care, lifting, headache, recreation work, driving, concentration, sleeping and reading. It is completed by patient related to different functional status. NDI is used with musculoskeletal (MSK) related neck pain, cervical radiculopathy and other cervical related problems. Each item is rated by choosing one of five response categories and transformed to a total score from 0 to 100 (worst possible).
Numeric Pain Rating Scale (NPRS) | 4th day
  Changes from the baseline, Numeric pain rating scale is used to measure the intensity of pain. Numeric pain rating scale is like Visual analogue scale, in which a straight line is drawn to tell the intensity of pain.1 to 10 is the range of NPRS in which 0 means no pain and 10 means the worst pain ever. The scoring is easy at NPRS and requires at least minimum of 1 minute to end.
Algometer | 4th day
  Changes from the Baseline, Algometer is a device for determining sensitiveness to pain caused by pressure. Pressure algometry is a valuable and reliable instrument in the assessment of MTrPs sensitivity. It has been used successfully for the evaluation of Myofascial Trigger Points (MTrPs), to confirm the diagnosis, and to quantify irritability. Therapeutic effectiveness of various procedures on MTrPs can be quantified by algometry
Goniometer: | 4th day
  Changes from the baseline, To measure the cervical Range of Motion (ROM's) a large plastic called Goniometer is used worldwide. In different clinical settings to measure ranges of extremities and spine Goniometer is used. For measuring cervical ROMs patient sits in upright posture with thoracic and lumbar spine stable with the chair. Knees and hip are at angle of 90/90 and feet stable on floor and arms on the sides of chair. Then patient is said to move the head in either positions as far as possible. Movements include extension, flexion, right or left side bending and rotation

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiarotto A, Clijsen R, Fernandez-de-Las-Penas C, Barbero M. Prevalence of Myofascial Trigger Points in Spinal Disorders: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2016 Feb;97(2):316-37. doi: 10.1016/j.apmr.2015.09.021. Epub 2015 Oct 17. PMID 26475933
- [Background] Vazquez-Delgado E, Cascos-Romero J, Gay-Escoda C. Myofascial pain syndrome associated with trigger points: a literature review. (I): Epidemiology, clinical treatment and etiopathogeny. Med Oral Patol Oral Cir Bucal. 2009 Oct 1;14(10):e494-8. doi: 10.4317/medoral.14.e494. PMID 19680218
- [Background] Fernandez-de-Las-Penas C, Simons D, Cuadrado ML, Pareja J. The role of myofascial trigger points in musculoskeletal pain syndromes of the head and neck. Curr Pain Headache Rep. 2007 Oct;11(5):365-72. doi: 10.1007/s11916-007-0219-z. PMID 17894927
- [Background] simons DG. Understanding effective treatments of myofascial trigger points. Journal of Bodywork and movement therapies. 2002;6(2):81-8.
- [Background] Saadat Z, Hemmati L, Pirouzi S, Ataollahi M, Ali-Mohammadi F. Effects of Integrated Neuromuscular Inhibition Technique on pain threshold and pain intensity in patients with upper trapezius trigger points. J Bodyw Mov Ther. 2018 Oct;22(4):937-940. doi: 10.1016/j.jbmt.2018.01.002. Epub 2018 Jan 17. PMID 30368338
- [Background] Ravichandran P, Ponni HK, Aseer PAL. Effectiveness of ischemic compression on trapezius myofascial trigger points in neck pain. International Journal of Physiotherapy. 2016;3(2):186-92.
- [Background] Lenehan KL, Fryer G, McLaughlin P. The effect of muscle energy technique on gross trunk range of motion. Journal of osteopathic medicine. 2003;6(1):13-8.
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hong C-Z. Algometry in evaluation of trigger points and referred pain. Journal of Musculoskeletal Pain. 1998;6(1):47-59.